CLINICAL TRIAL: NCT01646827
Title: An Open-label, Randomized, Parallel Arm, Bioavailability Trial of Aripiprazole IM Depot Administered in the Deltoid or Gluteal Muscle in Adult Subjects With Schizophrenia
Brief Title: An Open Label Study of Aripiprazole Intramuscular Injection in Subjects With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 31-11-290
Record Dates: First submitted 2012-06-18; First posted 2012-07-20 (Estimated); Results first posted 2014-07-31 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Schizophrenia
Keywords: Schizophrenia, extended release antipsychotic
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deltoid (Experimental): Deltoid injection site
  Interventions: Drug: Aripiprazole IM Depot
- Gluteal (Experimental): Gluteal injection site
  Interventions: Drug: Aripiprazole IM Depot

INTERVENTIONS:
Drug: Aripiprazole IM Depot — One injection of 400 mg aripiprazole IM depot
  Other Names: Abilify

SUMMARY:
The purpose of this study is to determine whether aripiprazole injection into the shoulder or the buttocks produces similar effects in the body

DETAILED DESCRIPTION:
Extended-release gluteal intramuscular (IM) injection of aripiprazole has been tested in subjects with schizophrenia for safety and tolerability. This study will compare the gluteal IM aripiprazole injection with deltoid IM aripiprazole injection for safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia
* Stabilized on oral antipsychotic medication
* Good physical health
* BMI 18 to 35 kg/m2
* Prior history of tolerating aripiprazole

Exclusion Criteria:

* Sexually active males who will not commit to utilizing 2 of the approved birth control methods or who will not remain abstinent during the trial and for 180 days following the last dose of trial medication, or have not had an orchidectomy or sexually active females of childbearing potential who will not commit to utilizing 2 of the approved birth control methods or who will not remain abstinent during the trial and for 150 days following the last dose of trial medication. Abstinence will be permitted if it is confirmed and documented at every trial visit. If employing birth control, 2 of the following precautions must be used: vasectomy, tubal ligation, vaginal diaphragm, intrauterine device, birth control pill, birth control depot injections, implant, condom or sponge with spermicide.
* Subjects who have met DSM-IV-TR criteria for substance abuse or dependence within the past 180 days; including alcohol and benzodiazepines, but excluding caffeine and nicotine.
* Subjects with a positive drug screen for cocaine or other drugs of abuse (excluding stimulants and other prescribed medications and marijuana).
* Use of any psychotropic medications other than their current antipsychotic medication.
* Use of any CYP2D6 and CYP3A4 inhibitors, or CYP3A4 inducers within 14 days (fluoxetine 28 days) prior to dosing and for the duration of the trial.
* Females who are pregnant or lactating.
* Subjects who had participated in a previous IM depot trial within the last one year; or who had previously enrolled and received trial medication in an aripiprazole IM depot clinical trial.
* Any major surgery within 30 days prior to enrollment.
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical, electrocardiographic, or clinical laboratory examinations.
* Subjects who have a significant risk of committing suicide based on history, routine psychiatric status examination, investigator's judgment, or who have an answer of "yes" on questions 4 or 5 (current or over the last 30 days) on the Baseline/Screening version of the Columbia Suicide Severity Rating Scale (C-SSRS).
* Subjects currently in an acute relapse of schizophrenia.
* Subjects with a current DSM-IV-TR diagnosis other than schizophrenia, including schizoaffective disorder, major depressive disorder, bipolar disorder, delirium, dementia, amnestic or other cognitive disorders. Also, subjects with borderline, paranoid, histrionic, schizotypal, schizoid or antisocial personality disorder.
* Subjects who were considered treatment-resistant to antipsychotic medication.
* Subjects who have had electroconvulsive therapy within 2 months of administration of trial drug.
* Subjects with a history of neuroleptic malignant syndrome or clinically significant tardive dyskinesia as assessed by the investigator.
* Any other sound medical reason not to be entered into the trial, as determined by the clinical investigator.
* Subjects who are known to be allergic, intolerant, or unresponsive to prior treatment with aripiprazole or other quinolinones.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2012-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Peters-Strickland, MD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (6):
- United States (6):
  - Comprehensive Clinical Development, Inc., Cerritos, California
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - CNRI - San Diego, San Diego, California
  - Neuropsychiatric Research Center of Orange County, Santa Ana, California
  - Comprehensive Clinical Development, Inc., Washington D.C., District of Columbia
  - Community Clinical Research, Inc., Austin, Texas

REFERENCES:
- [Derived] Raoufinia A, Peters-Strickland T, Nylander AG, Baker RA, Eramo A, Jin N, Bricmont P, Repella J, McQuade RD, Hertel P, Larsen F. Aripiprazole Once-Monthly 400 mg: Comparison of Pharmacokinetics, Tolerability, and Safety of Deltoid Versus Gluteal Administration. Int J Neuropsychopharmacol. 2017 Apr 1;20(4):295-304. doi: 10.1093/ijnp/pyw116. PMID 28204607

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This report presents results of a study on 37 adults with schizophrenia, conducted at 6 centers in the United States.
Pre-assignment Details: Participants were randomized 1:1 to receive a single dose of aripiprazole intramuscular (IM) depot (400 mg) in either the deltoid muscle or gluteal muscle according to the randomization schedule.
Groups:
- Aripiprazole IM Depot 400 mg: Deltoid: The participants in this group received single dose of aripiprazole IM depot (400 mg) injection in the deltoid muscle.
- Aripiprazole IM Depot 400 mg: Gluteal: The participants in this group received single dose of aripiprazole IM depot (400 mg) injection in the gluteal muscle.
Period: Overall Study
Arm/Group | Aripiprazole IM Depot 400 mg: Deltoid | Aripiprazole IM Depot 400 mg: Gluteal
Started | 18 | 19
Completed | 16 | 14
Not Completed | 2 | 5
Not completed — Lost to Follow-up | 0 | 3
Not completed — Physician Decision | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole IM Depot 400 mg: Deltoid | Aripiprazole IM Depot 400 mg: Gluteal | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.1 (11.0) | 45.9 (7.3) | 44.5 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 12 | 15 | 27

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Aripriprazole
Description: Relative bioavailability (Frel) of aripiprazole intramuscular (IM) depot injected in the deltoid muscle compared to the gluteal muscle based on aripiprazole maximum (peak) plasma concentrations (Cmax) PK parameter.
Time Frame: Day 1: 4 hr, 8 hr, and 12 hr post dose, Days 2, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 25, 28, 35, 42, 49, 56, 63, 70, 77, 84, 98, 112 and 126/Early termination
Population: The dataset for the PK analysis consisted of all dosed subjects who had evaluable aripiprazole and dehydro-aripiprazole PK parameters.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Aripiprazole IM Depot 400 mg: Deltoid | Aripiprazole IM Depot 400 mg: Gluteal
Number analyzed (Participants) | 16 | 17
ng/mL | 170 (58.6) | 136 (70.3)

2. Primary Outcome: Area Under the Concentration-Time Curve Infinity (AUC Infinity); Area Under the Concentration-Time Curve 28 (AUC 28), and Area Under the Concentration-Time Curve t (AUC t): Aripiprazole
Description: Relative bioavailability (Frel) of aripiprazole IM depot injected in the deltoid muscle compared to the gluteal muscle based on area under the concentration-time curve (AUC) from time zero to the time of last measurable concentration (AUCt), AUC time curve 28, and AUC from time zero to infinity PK parameters.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng day/mL
Arm/Group | Aripiprazole IM Depot 400 mg: Deltoid | Aripiprazole IM Depot 400 mg: Gluteal
Number analyzed (Participants) | 16 | 17
ng day/mL
  AUC infinity (n=16,14) | 7590 (2590) | 7920 (2580)
  AUC 28 (n=16,17) | 3120 (1150) | 2380 (1410)
  AUC t (n=16,17) | 7360 (2420) | 7340 (2360)

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Dehydro-Aripiprazole
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Aripiprazole IM Depot 400 mg: Deltoid | Aripiprazole IM Depot 400 mg: Gluteal
Number analyzed (Participants) | 16 | 17
ng/mL | 51.7 (23.3) | 34.6 (13.2)

4. Primary Outcome: Area Under the Concentration-Time Curve Infinity (AUC Infinity); Area Under the Concentration-Time Curve 28 (AUC 28), and Area Under the Concentration-Time Curve t (AUC t): Dehydro-Aripiprazole
Description: Relative bioavailability (Frel) of aripiprazole IM depot injected in the deltoid muscle compared to the gluteal muscle based on area under the concentration-time curve (AUC) from time zero to the time of last measurable concentration (AUCt), AUC time curve 28 and AUC from time zero to infinity PK parameters.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng day/mL
Arm/Group | Aripiprazole IM Depot 400 mg: Deltoid | Aripiprazole IM Depot 400 mg: Gluteal
Number analyzed (Participants) | 16 | 17
ng day/mL
  AUC infinity (n=16,14) | 2520 (836) | 2230 (630)
  AUC 28 (n=16,17) | 886 (445) | 538 (305)
  AUC t (n=16,17) | 2420 (805) | 1990 (603)

5. Secondary Outcome: Number of Participants Reporting Treatment Emergent Adverse Events (TEAE).
Description: Safety was measured according to standard adverse event collection as described in the adverse event section of the results.
Time Frame: Starting at the time the ICF was signed to Day 126/Early termination
Population: Population included all randomized participants who received at least one dose of drug, regardless of any protocol violation.
Measure: Number; unit: Participants
Arm/Group | Aripiprazole IM Depot 400 mg: Deltoid | Aripiprazole IM Depot 400 mg: Gluteal
Number analyzed (Participants) | 17 | 18
Participants
  Subjects with TEAEs | 14 | 18
  Subjects with serious TEAEs | 0 | 0
  Subjects with severe TEAEs | 1 | 1

6. Secondary Outcome: Number of Participants With Laboratory Values of Potential Clinical Relevance.
Description: The laboratory tests were collected and processed in accordance with directions from the clinical chemistry laboratory. Based on criteria for identifying laboratory values of potential clinical relevance, the abnormal values were noted. Some of the criteria are as follows: For fasting triglycerides: men: ≥ 160 mg/dL and women: ≥ 120 mg/dL; Fasting glucose: ≥ 115 mg/dL; Prolactin: > upper limit of normal (ULN); Neutrophils: ≤ 1,500/mm3; and Creatine phosphokinase: ≥ 3 x ULN.
Time Frame: Day 1, Day 28, Day 126/Early termination
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Aripiprazole IM Depot 400 mg: Deltoid | Aripiprazole IM Depot 400 mg: Gluteal
Number analyzed (Participants) | 17 | 18
Participants
  High fasting triglycerides (n=9,11) | 3 | 5
  High fasting glucose (n=9,11) | 3 | 0
  High prolactin (n=17,18) | 3 | 3
  Low absolute neutrophils (n=17,18) | 1 | 2
  High creatine phosphokinase (n=17,18) | 2 | 0

7. Secondary Outcome: Number of Participants With Vital Signs of Potential Clinical Relevance-Blood Pressure
Description: Vital sign assessment included orthostatic (supine and standing) blood pressure. Orthostatic assessments were made after participants had been in the supine position for at least 5 minutes and again after participants had been standing for 2 minutes, but not more than 3 minutes. Orthostatic hypotension defined as >/= 20 mm Hg decrease in systolic blood pressure and >/= 25 beats per minute increase in heart rate from supine to standing.
Time Frame: Day 1, Day 14, Day 28 and Day 126/Early termination
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Aripiprazole IM Depot 400 mg: Deltoid | Aripiprazole IM Depot 400 mg: Gluteal
Number analyzed (Participants) | 17 | 18
Participants
  Increase >/=15 mmHg in diastolic standing BP | 0 | 1
  Orthostatic hypotension | 0 | 0

8. Secondary Outcome: Number of Participants With Vital Signs of Potential Clinical Relevance-Temperature
Description: Vital sign assessment included body temperature measured in centigrade(C). Temperatures >=37.8°C and increase of >= 1.1°C were recorded.
Time Frame: Day 1, Day 14, Day 28 and Day 126/Early termination
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Aripiprazole IM Depot 400 mg: Deltoid | Aripiprazole IM Depot 400 mg: Gluteal
Number analyzed (Participants) | 17 | 18
Participants | 0 | 0

9. Secondary Outcome: Number of Participants With Vital Signs of Potential Clinical Relevance-Heart Rate
Description: Vital sign assessment included heart rate (supine and standing). Heart rate with increase or decrease of >/= 15 beats per minute were recorded.
Time Frame: Day 1, Day 14, Day 28 and Day 126/Early termination
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Aripiprazole IM Depot 400 mg: Deltoid | Aripiprazole IM Depot 400 mg: Gluteal
Number analyzed (Participants) | 17 | 18
Participants
  Heart rate: Supine: increase | 0 | 0
  Heart rate: Supine: decrease | 0 | 0
  Heart rate: Standing: increase | 0 | 0
  Heart rate: Standing: decrease | 0 | 0

10. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Measurements of Potential Clinical Relevance
Description: Three 12 lead ECGs were performed approximately 5 minutes apart at each time point. The participant were supine and at rest (for at least 10 minutes) prior to the first ECG and will remain supine through the final ECG. Based on criteria for identifying ECG measurements of potential clinical relevance, the abnormal values were noted. Some of the criteria are as follows: For bradycardia: ≤ 50 beats per minute (bpm); and for increase in QTc: QTc ≥ 450msec.
Time Frame: Day 1, Day 14, Day 28 and Day 126/Early termination
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Aripiprazole IM Depot 400 mg: Deltoid | Aripiprazole IM Depot 400 mg: Gluteal
Number analyzed (Participants) | 17 | 18
Participants
  premature ventricular contractions | 2 | 1
  T-wave inversions | 2 | 2
  Bradycardia and sinus bradycardia | 0 | 1
  Abnormalities in QTc intervals | 0 | 0

11. Secondary Outcome: Visual Analog Scale (VAS) Score at Day 1, Day 14, Day 28 and Last Visit.
Description: Injection site pain was assessed using a VAS, which was completed by the trial participant, and the investigator's assessment of most recent injection site, which was completed by the investigator. VAS is 100 mm line, 0=no pain, 100=unbearably painful.
Time Frame: Day 1, Day 14, Day 28 and last visit
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400 mg: Deltoid | Aripiprazole IM Depot 400 mg: Gluteal
Number analyzed (Participants) | 17 | 18
Units on a scale
  Day 1: 0.5 hour pre-dose (n=17, 18) | 1.2 (3.4) | 0.8 (1.6)
  Day 1: 1 hour post-dose (n=17, 18) | 3.1 (7.3) | 1.7 (2.7)
  Day 14 (n=16, 18) | 1.3 (3.7) | 0.3 (0.8)
  Day 28 (n=16, 18) | 0.5 (1.1) | 0.5 (1.3)
  Last visit (n=17, 18) | 2.2 (7.2) | 0.5 (1.3)

12. Secondary Outcome: Number of Participants With Categorical Scores on the Columbia Suicide Severity Rating Scale.
Description: This scale consists of a baseline evaluation that assesses the lifetime experience of the participant with suicide events and suicidal ideation and a post baseline evaluation that focuses on suicidality since the last trial visit.
Time Frame: Screening, Baseline, Week 1, Week 2, Week 8, Week 18 visit and Last visit.
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Aripiprazole IM Depot 400 mg: Deltoid | Aripiprazole IM Depot 400 mg: Gluteal
Number analyzed (Participants) | 17 | 18
Participants
  Screening: Suicidality (n=17,18) | 4 | 7
  Screening: Suicidal behaviour (n=17,18) | 2 | 5
  Screening: Suicidal ideation (n=17,18) | 4 | 7
  Baseline: Suicidality (n=17,18) | 0 | 0
  Baseline: Suicidal behaviour (n=17,18) | 0 | 0
  Baseline: Suicidal ideation (n=17,18) | 0 | 0
  Week 1: Suicidality (n=17,18) | 0 | 0
  Week 1: Suicidal behaviour (n=17,18) | 0 | 0
  Week 1: Suicidal ideation (n=17,18) | 0 | 0
  Week 2: Suicidality (n=16,18) | 0 | 0
  Week 2: Suicidal behaviour (n=16,18) | 0 | 0
  Week 2: Suicidal ideation (n=16,18) | 0 | 0
  Week 8: Suicidality (n=16,18) | 0 | 0
  Week 8: Suicidal behaviour (n=16,18) | 0 | 0
  Week 8: Suicidal ideation (n=16,18) | 0 | 0
  Week 18: Suicidality (n=16,14) | 0 | 0
  Week 18: Suicidal behaviour (n=16,14) | 0 | 0
  Week 18: Suicidal ideation (n=16,14) | 0 | 0
  Last visit: Suicidality (n=17,18) | 0 | 0
  Last visit: Suicidal behaviour (n=17,18) | 0 | 0
  Last visit: Suicidal ideation (n=17,18) | 0 | 0

ADVERSE EVENTS:
Time Frame: Events were recorded starting at the time the ICF is signed up to 125 days after the study drug administration.
Description: All randomized participants who received at least one dose of study drug (aripiprazole IM depot 400 mg), regardless of any protocol violation were included in the safety analysis.
Groups:
- Aripiprazole IM Depot 400 mg: Deltoid: The participants in this group received single aripiprazole IM depot (400 mg) injection in the deltoid muscle.
- Aripiprazole IM Depot 400 mg: Gluteal: The participants in this group received single aripiprazole IM depot (400 mg) injection in the gluteal muscle.
Arm/Group | Aripiprazole IM Depot 400 mg: Deltoid | Aripiprazole IM Depot 400 mg: Gluteal
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 14/17 | 18/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole IM Depot 400 mg: Deltoid (N=17) | Aripiprazole IM Depot 400 mg: Gluteal (N=18)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Gingival pain (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Axillary pain (General disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Injection site pain (General disorders) | 6 | 5
Injection site rash (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Furuncle (Infections and infestations) | 0 | 1
Hordeolum (Infections and infestations) | 0 | 1
Infected bites (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 0
Blood glucose increased (Investigations) | 1 | 0
Blood triglycerides increased (Investigations) | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 1 | 0
Glucose urine present (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Akathisia (Nervous system disorders) | 3 | 3
Dizziness (Nervous system disorders) | 0 | 3
Dyskinesia (Nervous system disorders) | 1 | 1
Dystonia (Nervous system disorders) | 1 | 1
Extrapyramidal disorder (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 4
Sedation (Nervous system disorders) | 1 | 2
Somnolence (Nervous system disorders) | 3 | 0
Tremor (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 1 | 1
Conversion disorder (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 2
Restlessness (Psychiatric disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is no agreement between PI and sponsor that restricts the PI's right to discuss or publish trial results after the trial is completed.